CLINICAL TRIAL: NCT03646032
Title: An mHealth Education Intervention for Encouraging STI Testing Uptake
Brief Title: Sexually Active Adolescent Focused Education
Acronym: SAAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benten Technologies, Inc. (Industry)
Collaborators: University of Alabama at Birmingham (Other); Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Tony Ma, President, Benten Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAAFE
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Health Risk Behaviors
Keywords: Mobile dating simulation game; Sexual education; HIV; STI; Consent
MeSH Terms: conditions — Health Risk Behaviors; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: A total of 200 AAA males and females will be recruited from Washington, DC (n=100) and Birmingham, Alabama (n=100). At both data collection sites, participants will be randomly assigned to one of two groups i.e., intervention and control during the pilot.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group (n=200) - will consist of 100 AAA males / 100 AAA females randomly selected participants who will receive a download of the SAAFE game and play for at least 30 minutes and as long as an hour, if desired.
  Interventions: Behavioral: SAAFE
- Control group (Active Comparator): Control group (n=200) - will consist of 100 AAA males / 100 AAA females randomly selected participants. This group will receive the standard of care by launching a mobile app that will play a dating sim game (called Choices). They will also receive pamphlets that provide information on the testing location and care if they have HIV/STI.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: SAAFE — After completing the pre-game assessment, participants will be asked to play the SAAFE game for at least 30 minutes and up to 1 hour . At the conclusion of the game, participants will be provided with a post-game assessment about their perception of risk, knowledge of specific protective behaviors, and whether they plan to change behaviors.
  Arms: Intervention group
Behavioral: Control — This group will receive dating sim game (called Choices). They will also receive pamphlets that provide information on the testing location and care if they have HIV/STI.
  Arms: Control group

SUMMARY:
SAAFE will be pilot tested in 2 geographically distinct areas (Washington, DC and Deep South) with 100 participants from each site to 1) primarily assess the efficacy of improved self-efficacy, knowledge about HIV/STIs and perception of sexual risks by AAAs, and (2) secondarily detect intention to be tested for STIs and to change sexual risk behavior (i.e., use a condom).

DETAILED DESCRIPTION:
A total of 200 African American adolescents (AAA) males and females will be recruited from Washington, DC (n=100) and Birmingham, Alabama (n=100). At both data collection sites, participants will be randomly assigned to one of two groups during the pilot. The two groups are:

1. Intervention group (n=100) - will consist of 50 AAA males / 50 AAA females randomly selected participants who will receive a download of the SAAFE game and play for at least 30 minutes and as long as an hour, if desired.
2. Control group (n=100) - will consist of 50 AAA males / 50 AAA females randomly selected participants. This group will receive dating sim game (called Choices). They will also receive pamphlets that provide information on the testing location and care if they have HIV/STI.

ELIGIBILITY:
Inclusion Criteria:

* African American female or male
* Between 15-21 years of age

Exclusion Criteria:

* Pregnant women
* The first 6 weeks post-partum
* Adolescents younger than 15

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 178 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Knowledge about HIV/STIs | 1 month
  During the pilot, adolescents will be asked if they would like to download the game to play on their own mobile device and complete a pre- and post-game assessment designed to measure their knowledge on HIV/STIs by assessing the level of knowledge around risky sexual activity.

SECONDARY OUTCOMES:
Perception of sexual risks | 1 month
  During the pilot, adolescents will be asked if they would like to download the game to play on their own mobile device and complete a pre- and post-game assessment designed to measure their perceived risk
Intention to be tested for STIs | 1 month
  We will ask participants on a scale of 1-5 their intent to get tested for HIV and most common STI's.
Intention to use a condom | 1 month
  We will ask participants on a scale of 1-5, their intent to use a condom.
Consent | 1 month
  We will ask participants on a 4-point Likert scale (strongly agree to strongly disagree)
System Usability and Acceptability Metrics | 1 month
  We will ask participants to answer the questions based on their current impressions on the game.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Ma, MS, Principal Investigator — Benten Technologies, Inc.
Locations (2):
- United States (2):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR, Analytic Code